CLINICAL TRIAL: NCT05199623
Title: The Effect of Chinese Herbal Medicine(Tailored Guizhi Decoction) as an Adjuvant Therapy in the Treatment of Traumatic Anosmia
Brief Title: The Effect of Chinese Herbal Medicine as an Adjuvant Therapy in the Treatment of Traumatic Anosmia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CF18227A
Record Dates: First submitted 2022-01-03; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Traumatic Anosmia
Keywords: Chinese herbal medicine; Guizhi decoction; Olfactory training; Phenyl ethyl alcohol threshold test; Traumatic anosmia; University of Pennsylvania Smell Identification Test
MeSH Terms: interventions — Olfactory Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHM(Chinese herbal medicine) group (Experimental): Treatment with steroid, zinc, and olfactory training for one month. And then, take CHM(Chinese herbal medicine) (tailored Guizhi decoction) and perform OT(olfactory training) for 6 months
  Interventions: Drug: tailored Guizhi decoction; Behavioral: Olfactory training (OT)
- OT(olfactory training) group (Active Comparator): Treatment with steroid, zinc, and olfactory training for one month. And then, perform OT(olfactory training) only for 6 months.
  Interventions: Behavioral: Olfactory training (OT)

INTERVENTIONS:
Drug: tailored Guizhi decoction — Tailored guizhi decoction powder is a compound Chinese herbal medicine which contains 7.0g of guizhi, 1.5g of chuanxiong, 1.5g of zhimu, 1.5g of xinyi, 0.3g of mahuang, 1.0g of baizh, 2.0g of jili, 1.5g of fuling, and 1.0g of danshen.
  Arms: CHM(Chinese herbal medicine) group
Behavioral: Olfactory training (OT) — Four odorant bottles of PEA, lemon, eucalyptus, and clove oils were given. Patients were instructed to sniff the liquid in each bottle for 10 seconds, twice a day.

SUMMARY:
Objective: To investigate the effect of Chinese herbal medicine (CHM) as an adjuvant therapy in the treatment of traumatic anosmia.

Methods: Patients with a clear history of loss of smell after head injury, and whose phenyl ethyl alcohol (PEA) odor detection threshold remained -1 after treatment with steroid, zinc, and olfactory training (OT) for one month, were included in this study between September of 2018 and November of 2020. They were randomly divided into 2 groups, with patients in the CHM group taking CHM (tailored Guizhi decoction) and performing OT, and those in the OT group receiving OT only for 6 months. After 3 months' and 6 months' treatment, the olfactory function was evaluated by both the PEA threshold test and the traditional Chinese version of the University of Pennsylvania Smell Identification Test (UPSIT-TC). Magnetic resonance imaging was performed to measure the volume of olfactory bulbs after 6 months' treatment.

ELIGIBILITY:
Inclusion Criteria:

* a clear history of loss of smell after an episode of head injury
* PEA threshold was -1, which is assumed to be anosmic

Exclusion Criteria:

* One month later, they received birhinal and unirhinal PEA threshold tests. Any patient whose birhinal or unirhinal threshold was below -1 was excluded from the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Olfactory test - Birhinal PEA threshold (3 months after treatment) | Change between before treatment and 3 months after treatment
  The PEA threshold test consists of different concentrations of a rose-like PEA odorant to measure the odor threshold. A 2-alternative forced-choice single-staircase procedure is used in the PEA test.
Olfactory test - Birhinal PEA threshold (6 months after treatment) | Change between before treatment and 6 months after treatment
  The PEA threshold test consists of different concentrations of a rose-like PEA odorant to measure the odor threshold. A 2-alternative forced-choice single-staircase procedure is used in the PEA test.
Olfactory test - UPSIT-TC (3 months after treatment) | Change between before treatment and 3 months after treatment
  UPSIT-TC is an odor identification test that is modified from the North American version of University of Pennsylvania Smell Identification Test(UPSIT). In the UPSIT-TC, 8 Odorants have been replaced to reflect the culture of the test-takers [20]. The UPSIT-TC is
  composed of 40 tests. In each test, an odorant is embedded in microcapsules and positioned on the brown bottom strips of the test page. The patient scratches the strip with a pencil tip to release the odorant. Then he or she sniffs the released odorant and chooses from a set of 4 odor descriptors to identify the odorant. The test is scored as the number of odors identified correctly
Olfactory test - UPSIT-TC (6 months after treatment) | Change between before treatment and 6 months after treatment
  UPSIT-TC is an odor identification test that is modified from the North American version of University of Pennsylvania Smell Identification Test(UPSIT). In the UPSIT-TC, 8 Odorants have been replaced to reflect the culture of the test-takers [20]. The UPSIT-TC is
  composed of 40 tests. In each test, an odorant is embedded in microcapsules and positioned on the brown bottom strips of the test page. The patient scratches the strip with a pencil tip to release the odorant. Then he or she sniffs the released odorant and chooses from a set of 4 odor descriptors to identify the odorant. The test is scored as the number of odors identified correctly
The volume of olfactory bulbs | 6 months after treatment
  MRI was performed to measure the volume of olfactory bulbs (OB) at the end of the treatment using a 1.5-Tesla Exite MRI system (GEMS, Milwaukee, WI, USA) with a quadrature head coil. The imaging pulse sequences included axial T1-weighted images, FLAIR images, along with axial and coronal T2-weighted fast spin-echo images. Contrast-enhanced T1-weighted images with axial and coronal sections were acquired. After a sagittal localizing scan, 2-2.5-mm-thick T2-weighted coronal and sagittal (both TR = 5,000 ms, TE = 106 ms, NEX = 2, Matrix = 256 9 256) images without an interslice gap were taken with a 12-cm field of view, as per the standardized protocol for OB analysis. OB volumes were measured using Mimics Medical 21.0 (Materialise, Leuven, Belgium).

CONTACTS AND LOCATIONS:
Overall Officials: Rong-San Jiang, Study Chair — Departments of Medical Research, Otolaryngology, Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No